CLINICAL TRIAL: NCT05293431
Title: Characterization and Modulation of Brain Networks to Promote Brain Resilience for the Coronavirus (COVID-19) Pandemic
Brief Title: Promote Brain Resilience for the Coronavirus (COVID-19) Pandemic
Acronym: MBNPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Guttmann (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Javier Solana Sanchez, PhD, Institut Guttmann
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021365
Record Dates: First submitted 2022-03-16; First posted 2022-03-24 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Transcranial Direct Current Stimulation; Mental Health Issue; Public Health; Resilience, Psychological; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Stimulation Group (Experimental): This group will receive real tACS non-invasive brain stimulation
  Interventions: Other: Transcranial Alternate Current Stimulation
- Sham Control Group (Sham Comparator): This group will receive Sham tACS non-invasive brain stimulation
  Interventions: Other: Sham stimulation

INTERVENTIONS:
Other: Transcranial Alternate Current Stimulation — tACS utilizes low-amplitude alternating currents to modulate brain activity and entrain specific brain oscillations depending on the applied stimulation frequency
  Arms: Active Stimulation Group
Other: Sham stimulation — Sham stimulation will simulated the real tACS stimulation
  Arms: Sham Control Group

SUMMARY:
Background:

By the end of 2020, the coronavirus disease (COVID-19) pandemic resulted in over 84 million cases and nearly 2 million deaths.

Continued confinement and restriction are expected to negatively affect mental health, however, some individuals are likely to show much less negative impact than others. The characterization and neurobiological determinants of brain resilience vs vulnerability during the pandemic should generate critical knowledge and open future avenues for individually tailored interventions.

Objectives:

1. Identify the individual psychobiological determinants of resilience during COVID-19 pandemic.
2. Conduct a non-invasive brain stimulation intervention to modulate the expression of resilience brain networks.

Methods:

Barcelona Brain Health Initiative participants will be included, encompassing multiple assessments before and during the COVID-19 pandemic. Machine learning techniques will be applied to define brain networks signature of resilience. Subsequently transcranial alternating stimulation will be used during a controlled trial intervention to promote the expression of brain resilience networks.

Expected results:

The present project should provide critical new knowledge on brain mechanisms underlying resilience and first evidences of the feasibility and impact of modulating brain resilience networks in terms of its effects on mental health of participants.

DETAILED DESCRIPTION:
As of the end of 2020, the coronavirus (COVID-19) pandemic had resulted in over 88 million confirmed cases and nearly 2 million deaths worldwide. Recurring waves of infection are forcing to impose continuing social restrictions and confinement measures all around the world.

From a public health perspective, these measures could potentially have an important negative impact on society and has led to the call for development of preventive and interventional strategies.

However despite the generalized negative effects of infection some individuals seem relatively protected from negative sequelae. Therefore, some people appear to be particularly resilient and the characterization and better understanding of characteristics that explain why some remain resilient has been highlighted as a critical focus of needed research, as it allows the potential to identify factors that can be targets for designing interventional strategies.

Resilience, the concept that describes the capacity of certain individuals to resist the impact of illness and distress, is a broad term. In clinical psychology and mental health, the concept of resilience has been historically been linked to the study of individual differences (e.g., self-esteem, sense of control, perception of social support, etc.) that determine the capacity to cope with the impact of life traumas in order to maintain normal psychological and physical functioning and avoid serious mental illness.

Beyond the psychological aspects, the determinants and factors that confer individual differences in resilience require integrated assessment of specific person's social context, engagement in positive lifestyles, and their interplay with its brain biological substrates and mechanisms. Neuroimaging investigations have identified brain regions that show specific activity and connectivity patterns during exposure to stressful or violent stimuli and that may be correlated with scores in psychosocial scales of resilience or predict subsequent coping abilities. Within the field of ageing and dementia some studies have suggested the role of the frontal cortex, specifically the functional connectivity of the dorsolateral prefrontal cortex to the rest of the brain or to particular networks (DMN, SN), as a neural substrate of higher resilience, both in normal aging.

A critical aspect to consider is that, while it is tempting to leverage such neuroimaging studies to try to identify a "human brain network of resilience", animal work on the neural substrate of resilience illustrates the importance of interventional experimental designs that employ stimuli that can be precisely quantified and controlled. Novel neuroscience approaches allow to undertake substantial translational work to enable the study of the neural substrates of resilience in humans, probing in a more direct causal association between brain circuit function and metrics of cognitive function or behavioral assessment - or subjective, i.e., related to wellbeing. As an example, the stress-response paradigm, offers a useful framework for the definition and study of resilience. It consists of three principal elements 1) a stressor; 2) an organism response; and 3) a given outcome.

Importantly, the experimental approach can also be applied to directly modulate the activity of brain networks subtending resilience processes.

Methods:

Can be actively modulate resilience? The main objective of subproject is to test the possibility to modulate the activity of the neural network underlying resilience and investigate the effects at the level of observable behavioral and neurophysiological changes.

Researchers propose a double-blind brain stimulation study.

Participants Participants will be pseudo-randomly selected, stratifying where possible for socio-demographical variables, amongst those individuals previously defined as "vulnerable".

Sample size was calculated considering the effect size of the few previous studies investigating the modulatory effect of non-invasive brain stimulation on functional and behavioral outcomes of resilience to stress previous studies of our group that showed how different non-invasive brain stimulation technique could differently modulate functional magnetic resonance (fMRI) derived brain networks dynamics or studies that employed stressor paradigms tasks to explore brain networks organization.

Non-invasive brain stimulation researchers will use transcranial alternating current stimulation (tACS), combined with neuroimaging data and high density EEG (hdEEG).

tACS utilizes low-amplitude alternating currents to modulate brain activity and entrain specific brain oscillations depending on the applied stimulation frequency. Researchers previously developed a method for optimizing the configuration of multifocal tACS for stimulation of specific brain networks (which effect can outlast the duration of stimulation and the use of a novel (sham) control stimulation paradigm will ensure the proper blinding of all participants.

tACS study protocol: general montage and configuration procedures tACS montages will be designed with the Stimweaver montage optimization algorithm to determine the positions and currents of the electrodes over the scalp that induce an electric field in the brain that better approximates a weighted target electric field map. Stimulation will be delivered using 8 circular electrodes with an area of 8 cm2. For safety issues, the maximum current delivered by any electrode will be 2 milliampere (mA), while the maximum current injected through all the electrodes will be 4 mA. In the real intervention conditions, the current will be supplied during the whole experimental session. In all groups, the current will be initially increased and finally decreased in a 30 s ramp-up and ramp-down fashion. For the sham condition, the current dosage will be composed of an initial ramp-up of 30 s immediately followed by a 1 min ramp- down, and a final ramp-down of 30 s immediately preceded by a ramp-up of 1 min. All stimulation parameters will adhere to general transcranial electrical stimulation current safety criteria guidelines.

Pre-post experimental stress coping paradigm To induce stress, researchers will use the moving-circles paradigm. In this task there are two circles moving sometimes closer and at times moving away from each other. When the circles touch, participants are delivered a mild electric stressor. Circle movement has a high degree of unpredictability and the circles might approach each other such that the stressor is more imminent, and then retreat from each other for a period.

Study design:

Double-blind controlled tACS study In order to evaluate the effect of stimulation on the modulation of the resilience networks, the researchers will implement a double-blind controlled trial using tACS.

Participants will receive tACS stimulation in two conditions which will be administered in a counterbalanced manner. In the first condition the researchers will target nodes of the resilience network identified by subproject#1, and in the second condition participants will receive sham stimulation. The study will be conducted in a double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

* No neurologic and neuropsychiatric diagnosis

Exclusion Criteria:

* Contraindication to receive safety tACS

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Resilience scale | The scale will be administered immediately before and immediately after the non invasive brain stimulation (up to 15/20) minutes
  Connor Davidson resilience scale (RISC-10)
Anxiety scale | The scale will be administered immediately before and immediately after the non invasive brain stimulation (up to 15/20) minutes
  State and Trait Anxiety Inventory the efficacy of the stimulations (STAI)
Stress scale | The scale will be administered immediately before and immediately after the non invasive brain stimulation (up to 15/20) minutes
  Holmes Stress Scale (HSS)
Stress scale | The scale will be administered immediately before and immediately after the non invasive brain stimulation (up to 15/20) minutes
  Acute Stress Appraisal questionnaire (ASA)
Heart Rate | During the execution of the stress inducing paradigm administered immediately before and immediately after the non invasive brain stimulation (up to 15/20) minutes
  During the stress inducing paradigm we will register heart rate variations
Pupillary response | During the execution of the stress inducing paradigm administered immediately before and immediately after the non invasive brain stimulation (up to 15/20) minutes
  During the stress inducing paradigm we will register variations in the diameter of the pupil
Skin conductance response | During the execution of the stress inducing paradigm administered immediately before and immediately after the non invasive brain stimulation (up to 15/20) minutes
  During the stress inducing paradigm we will register variations in the diameter of the pupil
EEG signal | During the execution of the stress inducing paradigm administered immediately before and immediately after the non invasive brain stimulation (up to 15/20) minutes
  We will explore changes in connectivity or oscillation of the network using EEG signal registered during the stress inducing task.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Guttmann, Badalona, Barcelona, Spain